CLINICAL TRIAL: NCT05388318
Title: Weight Reduction and Cognitive Health: A Remote Randomized Controlled Pilot Study Testing a Prolonged Nightly Fasting Intervention Among Obese, Stressed Mid-life Adults
Brief Title: Weight Reduction and Cognitive Health: Pilot Study Testing a Prolonged Testing Prolonged Fasting Among Obese, Stressed Mid-life Adults
Acronym: GetSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00015014
Record Dates: First submitted 2022-04-19; First posted 2022-05-24 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Midlife Obese Adults With Cognitive Decline

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 groups (intervention and control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged nightly fasting (PNF) (Experimental)
  Interventions: Behavioral: Prolonged nightly fasting
- Health Education Control (HEC) (Active Comparator)
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Prolonged nightly fasting — 14 hour nightly fast from caloric food and beverage; followed by 10 hour eating window. 8-week intervention duration.
  Arms: Prolonged nightly fasting (PNF)
Behavioral: Health Education Control — Weekly health education video viewing related to general health topics
  Arms: Health Education Control (HEC)

SUMMARY:
Using a randomized controlled trial (RCT) design, we will test feasibility and outcomes following an remotely delivered, nationwide 8-week prolonged nightly fasting (PNF) intervention compared to an health education control (HEC) in 50 obese, stressed mid-life adults to explore outcomes related to cognitive function, metabolism and associated lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 40-59 years old
* experiencing memory loss
* BMI 30-45.9
* PSS-4 score ≥5
* access to smartphone, zoom, and wifi
* lives in United States

Exclusion Criteria:

* diabetes
* pregnant,
* neurological disorder
* eating disorder within last 20 years
* In current weight loss program
* previously had bariatric surgery
* works a night shit
* health condition not conducive to nightly fasting

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Telephone Montreal Cognitive Assessment | 8 weeks
  T-MoCA, a measure of cognitive function
Every Day Cognition-12 | 8 weeks
  ECOG-12, a measure of cognitive function

SECONDARY OUTCOMES:
Perceived Stress Scale- 10 | 8 weeks
  PSS-10, a measure of perceived stress
Rapid Eating Assessment for Participants | 8 weeks
  REAPS, a measure of eating behaviors
Creature of Habit Scale | 8 weeks
  COHS, a measure of habitual behavior
Three-Factor Eating Questionnaire-Revised | 8 weeks
  TFEQ, a measure of eating behaviors
Pittsburgh Sleep Quality Index | 8 weeks
  PSQI, a measure of sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided